CLINICAL TRIAL: NCT04667884
Title: Effects of Prebiotic or Probiotic Supplements on Symptoms of Functional Constipation Among Adults
Brief Title: Effects of Prebiotic or Probiotic Supplements on Symptoms of Functional Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Jiaomei Yang, Assistant Professor, Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201911143
Record Dates: First submitted 2020-08-07; First posted 2020-12-16 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — Prebiotics; Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group A (Experimental): a mixture of Xylooligosaccharides, Stachyose, Fructooligosaccharides, and Water-soluble Dietary Fiber, 12 g/d, 4 weeks
  Interventions: Dietary Supplement: Prebiotics or Probiotics
- Group B (Experimental): a mixture of Fructooligosaccharide, water-soluble dietary fiber, polydextrose, and isomalt oligosaccharide, 12 g/d, 4 weeks
  Interventions: Dietary Supplement: Prebiotics or Probiotics
- Group C (Experimental): a mixture of Polydextrose, wheat fiber, and Seed shell of Plantago rotundifolia, 12 g/d, 4 weeks
  Interventions: Dietary Supplement: Prebiotics or Probiotics
- Group D (Experimental): a mixture of Fructooligosaccharides, Bifidobacterium lactis HN019 and Lactobacillus rhamnosus HN001, 3 g/d, 4 weeks
  Interventions: Dietary Supplement: Prebiotics or Probiotics
- Group E (Placebo Comparator): Maltodextrin， 3 g/d, 4 weeks
  Interventions: Dietary Supplement: Prebiotics or Probiotics

INTERVENTIONS:
Dietary Supplement: Prebiotics or Probiotics — All the supplements were provided in solid drinks，and required to drink with plain water 35-40℃, and lifestyle intervention was provided to all the groups by reading materials.

SUMMARY:
This study intends to evaluate the effects of three prebiotic solid beverages (mainly dietary fiber and prebiotics) and one probiotic solid beverage on the laxative effect of patients with functional constipation through randomized controlled trials. The influence of tract flora is expected to provide a basis for related therapies for patients with functional constipation.

ELIGIBILITY:
Inclusion Criteria:

1. Adults: 18 to 70 years old (not less than 50% of the final population over 45 years old, and not less than 30% of men);
2. Patients with functional constipation (refer to Rome IV diagnostic criteria for functional constipation); * Symptoms appeared for at least 6 months before diagnosis, and met the above diagnostic criteria in the past 3 months

Exclusion Criteria:

1. Pregnant and lactating women;
2. Unable to take the test sample and complete the inspection items as required due to inability to take food by mouth, weakness, allergies or other reasons (including the inability to complete all items due to recent travel plans);
3. Unclear main complaint and obvious abnormal mental state;
4. The liver and kidney function indexes are obviously abnormal (combined with the results of physical examination within the past 1 year);
5. Acute gastrointestinal diseases occurred in the past month, and constipation caused by surgical operations in the past month;
6. Take antibiotics, laxatives or topical agents, anticholinergics, antidiarrheals frequently in the past 1 month, and the frequency is more than 1 time/week
7. Have been diagnosed with the following diseases: cancer (especially cancer of the digestive tract), severe enteritis, intestinal obstruction, inflammatory bowel disease, hypothyroidism, mental illness;
8. Have been diagnosed with the following diseases: severe systemic diseases such as stroke, heart disease, liver cirrhosis, renal failure, hematopoietic system, or qualitative intestinal diseases caused by colonoscopy or imaging display;
9. In the past 3 months, there are often abdominal pain, abdominal pain accompanied by changes in bowel characteristics or frequency, blood in the stool, diarrhea or involuntary weight loss;
10. Clinical manifestations or diseases that other researchers believe are not suitable for participating in the project.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-05-22 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Number of bowel movements per week | week 0 to 4
  bowel movements will be recorded per week

SECONDARY OUTCOMES:
Classification of bowel status | day 0, 14, 28
  Classification according to the difficulty of defecation 9/5000 According to the difficulty of defecation
Bristol classification of stool characteristics | day 0, 14, 28
  Bristol classification
glucose | day 0, 14, 28
  Fasting plasma
HDL-C | day 0, 14, 28
  Fasting plasma
LDL-C | day 0, 14, 28
  Fasting plasma
TG | day 0, 14, 28
  Fasting plasma
Tch | day 0, 14, 28
  Fasting plasma
diversity and abundance of intestinal flora | day 0, 14, 28
  16s rRNA

CONTACTS AND LOCATIONS:
Overall Officials: Xin Liu, Principal Investigator — Xi'an Jiaotong University
Locations (1):
- Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lai H, Li Y, He Y, Chen F, Mi B, Li J, Xie J, Ma G, Yang J, Xu K, Liao X, Yin Y, Liang J, Kong L, Wang X, Li Z, Shen Y, Dang S, Zhang L, Wu Q, Zeng L, Shi L, Zhang X, Tian T, Liu X. Effects of dietary fibers or probiotics on functional constipation symptoms and roles of gut microbiota: a double-blinded randomized placebo trial. Gut Microbes. 2023 Jan-Dec;15(1):2197837. doi: 10.1080/19490976.2023.2197837. PMID 37078654